CLINICAL TRIAL: NCT06525402
Title: The Effect of Sodium Bicarbonate, Saline and Black Mulberry Syrup on The Degree of Oral Mucositis in Children Receiving Chemotherapy: A Randomized Controlled Trial
Brief Title: Effect of Sodium Bicarbonate, Saline and Black Mulberry Syrup on Degree of Oral Mucositis in Children Receiving Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Selda Ateş Beşirik, Assistant Professor, Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022/73
Record Dates: First submitted 2024-03-29; First posted 2024-07-29 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Oral Mucositis; Chemotherapy Effect
Keywords: Sodium Bicarbonate; Saline; Black Mulberry Syrup; Oral Mucositis; Chemotherapy; Children
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a randomized controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sodium Bicarbonate Group (Usual care) (Placebo Comparator): General routine oral care. In the clinic where the research was conducted, a guideline is routinely applied for the care of oral mucositis in line with the stages of oral mucositis. Sodium bicarbonate is used in line with this guideline. The first group will receive routine oral care in the clinic with sodium bicarbonate. It will be applied as a 5 ml mouthwash four times a day, after meals and before going to bed at night.
  Interventions: Other: Sodium Bicarbonate Group (Usual care)
- Saline Group (Experimental): It will be applied as a 5 ml mouthwash four times a day, after meals and before going to bed at night.
  Interventions: Other: Saline Group
- Black Mulberry Syrup Group (Experimental): It will be applied as a 5 ml mouthwash four times a day, after meals and before going to bed at night.
  Interventions: Other: Black Mulberry Syrup Group

INTERVENTIONS:
Other: Sodium Bicarbonate Group (Usual care) — In the clinic where the research was conducted, a guideline is routinely applied for the care of oral mucositis in line with the stages of oral mucositis. Sodium bicarbonate is used in line with this guideline. The first group, the control group, will receive routine oral care in the clinic with sodium bicarbonate. Oral care will be applied 4 times a day for 14 days.
  Arms: Sodium Bicarbonate Group (Usual care)
Other: Saline Group — The second group, the experimental group, will first receive oral care routinely applied in the clinic. Then, oral care will be given in the form of 5 ml mouthwash with saline. Oral care will be applied 4 times a day for 14 days.
  Arms: Saline Group
Other: Black Mulberry Syrup Group — The third group, the experimental group, will first receive oral care routinely applied in the clinic. Then black mulberry syrup will be applied. Then, oral care will be given in the form of 5 ml mouthwash with black mulberry syrup. Oral care will be applied 4 times a day for 14 days.
  Arms: Black Mulberry Syrup Group

SUMMARY:
This study was planned as a randomized controlled experimental study in order to compare the effects of oral care with saline and black mulberry syrup in addition to sodium bicarbonate on oral mucositis level in children aged 6-18 years receiving chemotherapy.

DETAILED DESCRIPTION:
Oral mucositis, also known as stomatitis, is the most common complication of cancer treatment. Mucositis affects the patient's nutrition, daily functions, and quality of life, may compromise the ability to tolerate scheduled therapy. For this reason, the children to be included in the study will be randomly divided into three groups. Sodium bicarbonate, which is the routine care in the clinic, will be administered to the control group, and to the intervention groups, saline in addition to the routine care and black mulberry syrup will be applied in addition to the routine care. Data will be collected according to Patient Information Form, International Child Mucositis Assessment Scale (ChIMES), World Health Organization Mucositis Classification and neutrophil counts. Oral care will be applied to the groups 4 times a day for 14 days. The International Child Mucositis Rating Scale (ChIMES), World Health Organization Mucositis Classification and neutrophil counts will be evaluated by the researchers on the 1st, 2nd, 4th, 8th and 16th days.

ELIGIBILITY:
Inclusion Criteria:

* The willingness of the family and the child to participate in the study
* Parent and child have separately informed written consent form
* Be between 6-18 years old
* Receiving chemotherapy and being hospitalized for chemotherapy treatment
* Being fed orally

Exclusion Criteria:

* Oral mucositis in the first intraoral evaluation
* Having diabetes
* Receiving radiotherapy
* Having a surgical procedure in the mouth and jaw area
* Receiving steroid therapy during chemotherapy treatment
* Using a method other than the methods used in the study to protect the oral mucous membrane throughout the study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Children's International Mucositis Evaluation Scale | up to 16 days
  Tomlison et al. (2010) developed Children's International Mucositis Evaluation Scale (ChIMES) in order to evaluate the difficulty experienced by children with cancer due to mouth/throat pain developing depending on mucositis. Yavuz et al., (2011) conducted the validity and reliability study of the Turkish version of the scale. The scale consists of six (6) questions and it is an easy-to-apply form that can be answered with the child's facial expressions.
Oral Mucositis Evaluation Index of the World Health Organization | up to 16 days
  It is scored between zero and four points. Although there is no change in the grade-0 mucosa, grade-1 painless ulcers, erythema or mild sensitivity, grade-2 painful erythema and ulcers, solid foods can be consumed. Grade-3 painful erythema, edema or ulcer can be consumed only, grade-4 ulceration, necrosis and hemorrhage are present, the patient cannot be fed, enteral or parenteral support is required.

SECONDARY OUTCOMES:
Neutrophil count | up to 16 days
  The neutrophil count will be evaluated. Numbers will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Selda Ateş Beşirik, Assistant Professor, Principal Investigator — Burdur Mehmet Akif Ersoy University
Locations (1):
- Isparta City Hospital, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No